CLINICAL TRIAL: NCT02794519
Title: 205076: A Phase II, Multicenter, Randomized, Double-blind (Sponsor-unblind), Placebo- Controlled, Parallel Group Trial to Evaluate the Efficacy and Safety of Sirukumab in Subjects With Severe, Poorly Controlled Asthma
Brief Title: A Phase 2a Study to Evaluate the Effects of Sirukumab in Subjects With Severe Poorly Controlled Asthma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This study has suspended participant recruitment.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205076
Record Dates: First submitted 2016-06-06; First posted 2016-06-09 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Asthma
Keywords: Asthma Control Questionnaire; interleukin-6; Sirukumab; severe, poorly controlled asthma; asthma; ACQ
MeSH Terms: conditions — Asthma | interventions — sirukumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sirukumab 50 mg/mL administered subcutaneously every 4 weeks (Experimental): Subjects will receive sirukumab 50 milligram/milliliter (mg/mL) subcutaneously every 4 weeks. They will receive the treatment for minimum of 20 weeks but up to 44 weeks of dosing. Sirukumab will be administered by the trained site staff at Baseline, Weeks 4 and Week 8. From the Week 12 visit onwards, subjects may start to self-administer study drug at the site under the supervision of the trained site staff if they are able and willing to do so. If not, study drug will continue to be administered by the trained site staff.
  Interventions: Drug: Sirukumab; Drug: Rescue medication
- Placebo administered subcutaneously every 4 weeks (Placebo Comparator): Subjects will receive placebo subcutaneously every 4 weeks. They will receive the treatment for minimum of 20 weeks but up to 44 weeks of dosing. Placebo will be administered by the trained site staff at Baseline, Weeks 4 and Week 8. From the Week 12 visit onwards, subjects may start to self-administer study drug at the site under the supervision of the trained site staff if they are able and willing to do so. If not, study drug will continue to be administered by the trained site staff.
  Interventions: Drug: Placebo; Drug: Rescue medication

INTERVENTIONS:
Drug: Sirukumab — This intervention will be provided in a 1.0 mL pre-filled syringe (PFS) fitted with spring-powered, disposable autoinjector device for single SC use that is permanently assembled on the syringe. The sirukumab PFS is aseptically filled to deliver a dose of 50 mg/1.0 mL of sirukumab.
  Arms: Sirukumab 50 mg/mL administered subcutaneously every 4 weeks
Drug: Placebo — This intervention will be provided in a 1.0 mL pre-filled syringe (PFS) fitted with spring-powered, disposable autoinjector device for single SC use that is permanently assembled on the syringe. The sirukumab PFS is aseptically filled to deliver a dose of 50 mg/1.0 mL of sirukumab.
  Arms: Placebo administered subcutaneously every 4 weeks
Drug: Rescue medication — Rescue medication (salbutamol/albuterol) shall be supplied to subjects at Screening for use when needed during the study.

SUMMARY:
Sirukumab is a fully human anti interleukin (IL)-6 immunoglobulin G1-kappa monoclonal antibody (MAb) which is in development for the treatment of rheumatoid arthritis (RA). The continuing unmet need in subjects with asthma refractory to corticosteroid therapy and increased understanding of asthma pathogenesis have stimulated the development of targeted biologics based on predictive biomarkers. The majority of approaches to date have targeted T Helper 2 (Th2) cytokines or their downstream effects. Targeting IL-6 in severe asthma represents an unprecedented approach that has potential to address non-Th2 drivers of severe asthma. This multicenter, randomized, double-blind (sponsor-unblind), placebo-controlled, parallel group study will investigate the efficacy of sirukumab compared to placebo in subjects having uncontrolled severe asthma despite use of high dose inhaled corticosteroid (ICS) in combination with long-acting Beta-agonist (LABA). The study will employ a variable treatment period for individual subjects. Dosing will continue every 4 weeks until week 44 (inclusive), or until 24 weeks after the final subject has been randomized, whichever the sooner. Upon receiving the final dose of study medicine or placebo, subjects will enter a 16 week Follow Up period. Overall, the duration of participation for subjects who complete the full 44-week treatment period and Follow Up period may be up to 64 weeks. Approximately 175 subjects will be randomized such that 140 evaluable subjects complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 - 75 years, inclusive.
* Severe, uncontrolled asthma according to the following criteria: Physician-diagnosed asthma for >=12 months, and; treatment for at least 3 months with >=880 microgram per day of fluticasone propionate (FP) dry powder for inhalation (DPI) or its equivalent, plus a long acting beta agonist (LABA), and' ACQ-7 score >=1.5, and; a documented history (e.g., medical record verification) in the 12 months prior to Visit 2 of >=1 exacerbation resulting in prescription for systemic oral corticosteroids or hospitalisation or extended observation in a hospital emergency room or outpatient centre. [For subjects on maintenance systemic corticosteroids, at least double the existing maintenance dose for at least 3 days is required] and; pre-bronchodilator FEV1 35-80% inclusive, with evidence of >=12% (and 200 milliliter [mL]) reversibility in FEV1 measured 15-30 minutes following 4 actuations of salbutamol (100 microgram per actuation) or albuterol (90 microgram per actuation) via pre-metered dose inhaler (pMDI). This reversibility criterion should have been documented in the 12-months prior to Screening. If no prior data are available this should be demonstrated either at Screening (Visit 2) or at the Randomization visit (Visit 3); blood eosinophil count <300 cells per microliter at screening.
* Body mass index 18-45 kilogram per meter square.
* Male or Females and Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until a cycle of spermatogenesis following five terminal half- lives after the last dose of study medication: Vasectomy with documentation of azoospermia; Male condom plus partner use of one of the following contraceptive options: Contraceptive subdermal implant; Intrauterine device or intrauterine system; Combined estrogen and progestogen oral contraceptive; Injectable progesterone; Contraceptive vaginal ring; Percutaneous contraceptive patches.
* This is an all-inclusive list of those methods that meet the following GlaxoSmithKline (GSK) definition of highly effective: having a failure rate of less than 1% per year when used consistently and correctly and, when applicable, in accordance with the product label. For non-product methods (e.g., male sterility), the investigator determines what is consistent and correct use. The GSK definition is based on the definition provided by The International Council for Harmonization of Technical Requirements for Pharmaceuticals for Human Use (ICH).
* The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
* A female subject is eligible to participate if she is of non-child bearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as age greater than 60 or 12 months of spontaneous amenorrhea with an appropriate clinical profile [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) >40 milliinternational units per milliliter (MlU/mL) and estradiol <40 picogram per milliliter (pg/mL) (<140 picomole per liter [pmol/L] is confirmatory) or if of child-bearing potential is using a highly effective method for avoidance of pregnancy for the duration of dosing and until 4 months post last-dose.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Presence of a known pre-existing, clinically important lung condition other than asthma. This includes chronic obstructive pulmonary disease (COPD), bronchiectasis, pulmonary fibrosis, bronchopulmonary aspergillosis, or a history of lung cancer.
* Lower respiratory tract infection (LRTI) or asthma exacerbation requiring antibiotics or systemic corticosteroids within 6 weeks of screening.
* Evidence of respiratory infection at screening.
* Has a history of chronic or recurrent infectious disease or ongoing infection including, but not limited to, chronic renal infection, chronic chest infection, recurrent urinary tract infection (example, recurrent pyelonephritis, chronic non-remitting cystitis), or open, draining skin wound or an ulcer.
* Serious infection within 8 weeks of enrolment, including, but not limited to hepatitis, pneumonia, sepsis, or pyelonephritis; or has been hospitalized for an infection; or has been treated with intravenous (IV) antibiotics for an infection, within 8 weeks prior to the first administration of study drug.
* Opportunistic infection, example, a nontuberculous mycobacterial infection or cytomegalovirus, pneumocystosis, aspergillosis within 6 months prior to screening.
* Evidence of poorly controlled chronic medical conditions other than asthma, example, subjects with known, pre-existing, clinically significant endocrine, autoimmune, metabolic, neurological, renal, gastrointestinal, hepatic, and haematological or any other system abnormalities that are uncontrolled with standard treatment.
* Current history of suicidal ideation or a past history of suicide attempt.
* Lactating, pregnant, or planning to become pregnant during the study.
* Malignancy within 5 years (except local basal cell carcinoma, or fully excised local dermal, squamous cell carcinoma).
* Has a history of known demyelinating diseases such as multiple sclerosis or optic neuritis.
* Has a history of gastrointestinal perforation or currently has active diverticulitis.
* QTcorrected (QTc) >450 milliseconds (msec) or QTc >480 msec in subjects with Bundle Branch Block. Notes: The QTc is the QT interval corrected for heart rate according to Bazett's formula (QTcB), Fridericia's formula (QTcF), and/or another method, machine-read or manually over-read; The specific formula that will be used to determine eligibility and discontinuation for an individual subject should be determined prior to initiation of the study. In other words, several different formulae cannot be used to calculate the QTc for an individual subject and then the lowest QTc value used to include or discontinue the subject from the trial.
* Alanine transaminase (ALT) >1.5 times upper limit of normal (ULN) and bilirubin >ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Laboratory abnormalities: Neutrophils <1.95 multiplied by 10 raise to 9 per liter; Platelet count <140 multiplied by 10 raise to 9 per liter; Hemoglobin <8.5 grams per decilitre (g/dL); WBC count <3.5 × multiplied by 10 raise to 9 per liter.
* Use of systemic corticosteroids within 6 weeks of screening. The only exception is subjects who take <=10 mg prednisolone (or equivalent) orally per day for chronic maintenance therapy, and who have been maintained on this regimen for >=12 weeks.
* The subject has received an investigational drug within 30 days or 5-half-lives (whichever is longer) prior to the first dose of study drug.
* Use of other monoclonal antibodies within 3 months (or 130 days in the case of Xolair) of screening.
* Live virus or bacterial vaccine from 30 days before screening.
* Immunomodulatory/suppressive agents including but not limited to cyclophosphamide, a cytotoxic agent, cyclosporine A, azathioprine, tacrolimus, mycophenolate mofetil, oral or parenteral gold, or D-penicillamine within 3 months of screening.
* Bronchial thermoplasty within 12 months of screening.
* Subjects with a smoking history of >=10 pack years (pack years = number of cigarettes smoked per day divided by 20 into number of years smoked). Note: Subjects who are current smokers, or ex-smokers (having given up smoking for >=6 months), are eligible for the study if their smoking history is <10 pack years.
* History of alcohol or illegal substance abuse consumption within 2 years of the study start.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation. Has any condition that, in the opinion of the investigator, would make participation not be in the best interest (example, compromise the well-being) of the subject or that could prevent, limit, or confound the protocol-specified assessments.
* Is an employee of the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, as well as family members of the employees or the investigator.
* Chest X-Ray (CXR) within 6 months of screening showing evidence of active or inactive tuberculosis (TB), or other clinically significant disease other than asthma. If a CXR is not available, it must be performed at screening.
* Positive for Mycobacterium tuberculosis using QuantiFERON Gold test at screening.
* Human Immunodeficiency Virus (HIV) positive or determined to be HIV positive at screening, testing to be conducted in accordance with local practice.
* Presence of hepatitis B surface antigen (HBsAg) or core antigen (HBcAg). Subjects who are HBsAg negative, but hepatitis core antigen positive may be included if they are polymerase chain reaction (PCR) negative for Hepatitis B deoxyribonucleic acid (DNA).
* Positive hepatitis C (Hep C) test result at screening or within 3 months prior to first dose of study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09-23 (Actual); Primary Completion 2016-10-04 (Actual); Study Completion 2016-10-04 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Asthma Control Questionnaire-7 (ACQ-7) at Week 24 | Baseline and Week 24
  The ACQ-7 is a seven-item questionnaire that is a measure of a subject's asthma control. Six of the questions will be self-completed by the subject, recalling over the previous 7 days. The six questions enquire about the frequency and/or severity of symptoms (nocturnal awakening, activity limitation, shortness of breath and wheeze), and rescue bronchodilator use. The response options for all these questions consist of a zero (no impairment/limitation) to six (total impairment/ limitation) scale. The final question is a rating of forced expiratory volume in 1 second FEV1% predicted. The questions are equally weighted and the ACQ score is the mean of the 7 questions and therefore between 0 (totally controlled) and 6 (severely uncontrolled). Baseline value is the value obtained at Day 1 before administration of investigational product (IP). Change from baseline in ACQ-7 score will be analysed using a Bayesian repeated measures model.

SECONDARY OUTCOMES:
Safety as assessed by number of subjects with adverse events (AE) and serious adverse events (SAE) | Up to 60 Weeks
  AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgement.
Safety as assessed by body temperature | Up to 60 Weeks
  Body temperature will be measured in semi-supine position after 5 minutes rest.
Safety as assessed by systolic and diastolic blood pressure | Up to 60 Weeks
  Blood pressure will be measured in semi-supine position after 5 minutes rest.
Safety as assessed by pulse rate | Up to 60 Weeks
  Pulse rate will be measured in semi-supine position after 5 minutes rest.
Safety as assessed by electrocardiogram (ECG) | Up to 60 Weeks
  Centralized 12-lead ECG will be performed in triplicate at baseline and singly thereafter. ECG will also be performed when clinically indicated. ECG measurements will be made after the subject has rested in the supine position for 5 minutes. The ECG will be obtained after the vital signs assessments but before lung function testing followed by other study procedures. Collection shortly after a meal or during sleep will be avoided since QT prolongation can occur at these times.
Safety as assessed by number of subjects with abnormal hematology parameters | Up to 48 Weeks
  Hematology will include hemoglobin, hematocrit, red blood cells (RBC) count, white blood cells (WBC) count, absolute neutrophils, neutrophils segmented percentage with differential, neutrophils bands percentage, basophils percentage, eosinophils percentage, absolute eosinophils, lymphocytes percentage, monocytes percentage, platelet count.
Safety assessed by serum chemistry | Up to 48 Weeks
  Serum chemistry will include potassium, chloride, sodium, calcium, blood Urea nitrogen (BUN), creatinine, glucose, aspartate transaminase (SGOT), alanine transaminase (SGPT), alkaline phosphatise, phosphate, albumin, total protein, direct, indirect and total bilirubin.
Safety assessed by lipid profile | Up to 48 Weeks
  Lipid profile will include total cholesterol, low density lipoprotein (LDL), high density lipoprotein (HDL), triglycerides.
Change from baseline in ACQ-7 during the treatment period | Baseline and Up to 48 Weeks
  The ACQ-7 is a seven-item questionnaire that is as a measure of a subject's asthma control.
Change from baseline in ACQ-5 during the treatment period | Baseline and Up to 48 Weeks
  The ACQ-5 is a five-item questionnaire that is as a measure of a subject's asthma control. The five ACQ-5 questions are scored on a 7-point scale (0 = good control, 7 = poor control), and the overall score is the mean of the five responses. Baseline value is the value obtained at Day 1 before administration of investigational product (IP). Change from baseline in ACQ-5 score will be analysed using a Bayesian repeated measures model.
Number of subjects who achieve an ACQ-7 response | Up to 48 Weeks
  The ACQ-7 is a seven-item questionnaire that is as a measure of a subject's asthma control.
Change from baseline in pre-bronchodilator FEV1 during the treatment period | Baseline and Up to 48 Weeks
  FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Baseline value is the value obtained at Day 1 before administration of IP. Change from Baseline is the difference between the value at Indicated visit and value at Baseline.
Change from baseline in average morning peak expiratory flow rate (PEFR) | Baseline and Up to 48 Weeks
  PEFR is the maximum flow rate generated during a forceful exhalation, starting from full lung inflation. Baseline value is the value obtained at Day 1 before administration of IP. Change from Baseline is the difference between the value at Indicated visit and value at Baseline.
Change from baseline in St. George's Respiratory Questionnaire (SGRQ) | Baseline and Up to 48 Weeks
  The SGRQ comprises 50 questions designed to measure health status (quality of life) in subjects with diseases of airways obstruction. The SGRQ includes a total score and three domain scores: Symptoms, Activity and Impacts (Psycho-social) as well as a total score. A minimum change in score of 4 units is considered to be established as clinically relevant. A one month recall period shall be used for assessment of the SGRQ. Baseline value is the value obtained at Day 1 before administration of IP. Change from Baseline is the difference between the value at Indicated visit and value at Baseline.
Number of subjects who achieve SGRQ response | Up to 48 Weeks
  The SGRQ comprises 50 questions designed to measure health status (quality of life) in subjects with diseases of airways obstruction.
Change from baseline in daily salbutamol/albuterol use | Baseline and Up to 48 Weeks
  Subjects will complete the Asthma Daily Symptom Diary (ADSD), a novel asthma symptom diary and record daily use of rescue medication (salbutamol/albuterol) via an electronic diary. Baseline value is the value obtained at Day 1 before administration of IP. Change from Baseline is the difference between the value at Indicated visit and value at Baseline.
Annualized rate of severe asthma exacerbations during the treatment period | Baseline and Up to 48 Weeks
  Severe asthma exacerbations are defined as worsening of asthma which requires use of systemic corticosteroids and/or hospitalisation and/or Emergency Department (ED) visits.
Assessment of pharmacokinetics (PK) of sirukumab | Blood sample for PK analysis would be collected at Baseline, Week 1, Week 4, Week 8, Week 12, Week 24, Week 48, Week 54 and Early Withdrawal/Week 60.
  Serum concentrations of sirukumab and derived population PK parameters will be evaluated. Blood samples for PK analyses of sirukumab serum concentrations will be drawn prior to the administration of study drug.
Change from baseline in blood or serum pharmacodynamic (PD) biomarkers including but not limited to interleukin (IL)-6 and C-reactive protein (CRP) | Blood sample for analysis of PD biomarkers would be collected at Baseline, Week 1, Week 4, Week 8, Week 12, Week 24, Week 48, Week 54 and Early Withdrawal/Week 60.
  Baseline value is the value obtained at Day 1 before administration of investigational product (IP). Change from Baseline is the difference between the value at Indicated visit and value at Baseline.
Incidence and titres of serum anti-sirukumab antibodies post-dosing | Blood sample for testing antibodies against sirukumab would be collected at Baseline, Week 12, Week 24, Week 48 and Early Withdrawal/Week 60.
  Analysis of anti-sirukumab antibodies will be performed using validated bioanalytical assays.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- United States (4):
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Richmond, Virginia
- Spain (3):
  - GSK Investigational Site, Alcorcón (Madrid)
  - GSK Investigational Site, Girona
  - GSK Investigational Site, Santiago de Compostela. La Coruña.